CLINICAL TRIAL: NCT00998998
Title: Iron Deficiency Anemia and Infant Behavior: Early Intervention Study II
Brief Title: The Anemia Control Program: Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Betsy Lozoff, MD, Professor of Pediatrics and Communicable Diseases and Research Professor, Center for Human Growth and Development, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD014122 (NIH)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-06

CONDITIONS: Iron Deficiency Anemia
Keywords: iron deficiency anemia; infant behavior; infant development
MeSH Terms: conditions — Anemia, Iron-Deficiency; Infant Behavior | interventions — Iron

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- 1 (Experimental): 6 or 12 month old infants with iron deficiency anemia assigned to receive home stimulation program via weekly home visits over 1 year
  Interventions: Behavioral: Home stimulation; Dietary Supplement: Iron
- 2 (Active Comparator): 6 or 12 month old infants with iron deficiency anemia assigned to surveillance (weekly visits to monitor health and iron supplement) over 1 year
  Interventions: Behavioral: Surveillance; Dietary Supplement: Iron
- 3 (Experimental): Nonanemic infants identified at 6 or 12 months assigned to receive home stimulation program via weekly home visits over 1 year
  Interventions: Behavioral: Home stimulation; Dietary Supplement: Iron
- 4 (Active Comparator): Nonanemic infants identified at 6 and 12 months assigned to surveillance (weekly visits to monitor health) over 1 year
  Interventions: Behavioral: Surveillance; Dietary Supplement: Iron

INTERVENTIONS:
Behavioral: Home stimulation — Weekly visit of one hour to the home over the course of one year to foster the mother-child relationship.
  Arms: 1; 3
Behavioral: Surveillance — Weekly visits to the home over the course of one year to record iron intake, feeding, and health information.
  Arms: 2; 4
Dietary Supplement: Iron — Six-month-old infants treated orally for 1 y with 15 mg elemental Fe/d as ferrous sulfate. Twelve-month old infants treated orally for a minimum of 6 months with 30 mg elemental Fe/d.

SUMMARY:
The purpose of this study was to determine if a home-based intervention to foster child development improved behavior and development in infants with IDA.

DETAILED DESCRIPTION:
Iron-deficiency anemia (IDA) is associated with alterations in infant behavior and development that may not correct with iron therapy. The purpose of this study was to determine if a home-based intervention to foster child development improved behavior and development in infants with IDA. IDA and non-anemic infants were randomly assigned to a year of intervention or surveillance only. Infants were enrolled and began study participation at 6 or 12 months. All infants were treated with oral iron and visited weekly to record iron intake, feeding, and health (surveillance). For infants randomized to intervention, the weekly home visit included an hour-long program fostering child development by supporting the mother-infant relationship. Psychologists, unaware of iron status or intervention assignment, assessed cognitive, motor, and social-emotional development (Bayley Scales) at the beginning, midpoint, and end of the year.

ELIGIBILITY:
Inclusion Criteria:

* birth weight >= 3.0kg
* singleton full-term birth
* routine vaginal delivery
* no major congenital anomalies
* no major perinatal complications
* no photo therapy
* no hospitalization for longer than 5 days
* no chronic illness
* no iron therapy
* from 1991-94, infants on >= 250 ml/day cow milk or formula
* from 1994-96, infants could be on < 250 ml/day cow milk or formula
* infants identified as anemic at 6 or 12 months and randomly selected nonanemic infants at 6 and 12 months

Exclusion Criteria:

* residence outside 4 contiguous working-class communities on outskirts of Santiago, Chile
* another infant <12 months in household
* infant in child care
* illiterate or psychotic caregiver or no stable caregiver available to accompany the child for appointments.
* until mid-1994, "exclusive" breastfeeding, defined as >250 mL/d cow milk or formula

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 277 (Actual)
Dates: Start 1992-04; Primary Completion 1996-07 (Actual); Study Completion 1996-07 (Actual)

PRIMARY OUTCOMES:
Infant behavior and development | 6, 12, and 18 months; or 12, 18, and 24 months

SECONDARY OUTCOMES:
Iron-deficiency anemia | 6, 12, and 18 months; or 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Lozoff, MD, Principal Investigator — University of Michigan
Locations (1):
- Instituto de Nutrición y Tecnología de los Alimentos (INTA), Santiago, Chile

REFERENCES:
- [Derived] Lozoff B, Smith JB, Clark KM, Perales CG, Rivera F, Castillo M. Home intervention improves cognitive and social-emotional scores in iron-deficient anemic infants. Pediatrics. 2010 Oct;126(4):e884-94. doi: 10.1542/peds.2009-3535. Epub 2010 Sep 20. PMID 20855384